CLINICAL TRIAL: NCT04497155
Title: The Association of Norepinephrine Use in Pre-hospital Transport and Early Mortality in Hemorrhagic Shock
Brief Title: Prehospital Norepinephrine and Early Mortality in Traumatic Shock
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Beaujon Hospital (Other); University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Justin Richards, Associate Professor of Anesthesiology, University of Maryland, Baltimore
Other Study IDs: HP-00082182
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Traumatic Shock; Hemorrhagic Shock; Traumatic Brain Injury; Hypotension and Shock
Keywords: hypotension; norepinephrine; traumatic shock
MeSH Terms: conditions — Shock, Traumatic; Shock, Hemorrhagic; Brain Injuries, Traumatic; Hypotension; Shock | interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prehospital norepinephrine: Trauma patients that received norepinephrine in the prehospital setting or in the resuscitation unit .
  Interventions: Drug: Norepinephrine
- Prehospital no norepinephrine: Trauma patients that did not receive norepinephrine in the prehospital setting or in the resuscitation unit.

INTERVENTIONS:
Drug: Norepinephrine — Trauma patients with prehospital or arrival to the trauma center hypotension, defined as a systolic blood pressure <100 mmHg, that received norepinephrine during prehospital transport or in the resuscitation unit.
  Groups: Prehospital norepinephrine

SUMMARY:
The effect of early, prehospital norepinephrine use in patients with traumatic shock on mortality is unknown. Recent existing observational evidence from single system data (US, France, Japan) are conflicting. The investigators hypothesize that prehospital norepinephrine is associated with decreased mortality when used in patients with traumatic shock.

DETAILED DESCRIPTION:
Prehospital hypotension is associated with worse clinical outcomes in patients who sustain traumatic injuries. Administration of vasoactive medications, including norepinephrine, is not advocated in North American trauma systems due to the belief that vasopressors will worsen clinical outcomes and increase mortality. However, in European trauma systems prehospital vasopressor administration is included as part of the guidelines for the management of hypotension and hemorrhagic shock. There are multiple physiologic explanations for why prehospital vasopressor administration may be useful in patients with traumatic shock, such as providing adequate blood pressure to maintain vital signs until arrival at the trauma center, allowing adequate organ perfusion in the setting of low blood flow, and supplementing decreased hormone production in the later stages of hemorrhagic shock.

The purpose of this retrospective study is to investigate if prehospital norepinephrine administration is associated with decreased mortality in patients with traumatic shock. The investigators will collect patient data from previously collected sources of information and trauma databases from three separate locations: the TRAUMABase consortium in Paris, France; TRENAU trauma database from Grenoble, France; and the R Adams Cowley Shock Trauma Center in Baltimore, MD, USA. The investigators will perform statistical modeling to propensity score match patients that received prehospital vasopressors with patients that did not receive prehospital vasopressors and assess the association with 24-hour and 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Blunt traumatic mechanism of injury
* Admitted to the trauma center from the scene of injury
* Systolic blood pressure during prehospital transport or at admission to the trauma center <100 mmHg

Exclusion Criteria:

* Penetrating mechanism of injury
* No vital signs at the scene of injury
* Prehospital cardiac arrest
* Transferred to the trauma center from another hospital

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be collected from the previously collected trauma database at three separate locations, as previously described. These databases are collected, maintained, and managed by professional medical staff.
Sampling Method: Non-Probability Sample
Enrollment: 2164 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Early mortality | Admission to the trauma center to 24-hours after admission
  Death within 24-hours of admission to the trauma center

SECONDARY OUTCOMES:
28-day mortality | Admission to the trauma center to 28-days after admission
  Death occurring within 28-days from admission to the trauma center

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Gauss, MD, Study Director — Hospital Beujon; Pierre Bouzat, MD, PhD, Study Director — University Grenoble Alps; Justin E Richards, MD, Principal Investigator — R Adams Cowley Shock Trauma Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta B, Garg N, Ramachandran R. Vasopressors: Do they have any role in hemorrhagic shock? J Anaesthesiol Clin Pharmacol. 2017 Jan-Mar;33(1):3-8. doi: 10.4103/0970-9185.202185. PMID 28413267
- [Background] Beloncle F, Meziani F, Lerolle N, Radermacher P, Asfar P. Does vasopressor therapy have an indication in hemorrhagic shock? Ann Intensive Care. 2013 May 22;3(1):13. doi: 10.1186/2110-5820-3-13. PMID 23697682
- [Result] Gauss T, Gayat E, Harrois A, Raux M, Follin A, Daban JL, Cook F, Hamada S; TraumaBase Group; Prehospital Traumabase Group Ile de France, SAMU=Service d'Aide Medicale Urgente. Effect of early use of noradrenaline on in-hospital mortality in haemorrhagic shock after major trauma: a propensity-score analysis. Br J Anaesth. 2018 Jun;120(6):1237-1244. doi: 10.1016/j.bja.2018.02.032. Epub 2018 Apr 14. PMID 29793591
- [Result] Sims CA, Holena D, Kim P, Pascual J, Smith B, Martin N, Seamon M, Shiroff A, Raza S, Kaplan L, Grill E, Zimmerman N, Mason C, Abella B, Reilly P. Effect of Low-Dose Supplementation of Arginine Vasopressin on Need for Blood Product Transfusions in Patients With Trauma and Hemorrhagic Shock: A Randomized Clinical Trial. JAMA Surg. 2019 Nov 1;154(11):994-1003. doi: 10.1001/jamasurg.2019.2884. PMID 31461138
- [Result] Harrois A, Baudry N, Huet O, Kato H, Dupic L, Lohez M, Ziol M, Vicaut E, Duranteau J. Norepinephrine Decreases Fluid Requirements and Blood Loss While Preserving Intestinal Villi Microcirculation during Fluid Resuscitation of Uncontrolled Hemorrhagic Shock in Mice. Anesthesiology. 2015 May;122(5):1093-102. doi: 10.1097/ALN.0000000000000639. PMID 25782753